CLINICAL TRIAL: NCT03482102
Title: A Phase II Trial of Durvalumab (MEDI4736) and Tremelimumab and Radiation Therapy in Hepatocellular Carcinoma and Biliary Tract Cancer
Brief Title: Durvalumab (MEDI4736) and Tremelimumab and Radiation Therapy in Hepatocellular Carcinoma and Biliary Tract Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Theodore Sunki Hong, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-517
Record Dates: First submitted 2018-03-14; First posted 2018-03-29 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Hepatocellular Carcinoma; Biliary Tract Cancer
Keywords: Hepatocellular Carcinoma; Biliary Tract Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Biliary Tract Neoplasms | interventions — tremelimumab; durvalumab; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tremelimumab + Durvalumab + Radiation (Experimental): * Durvalumab via IV infusion every 28 days for up to 4 doses/cycles
  * Tremelimumab via IV infusion every 28 days for up to 4 doses/cycles, and then continue durvalumab monotherapy every 4 weeks starting on Week 16 for up to 8 months.
  * Radiation therapy will only be given during cycle 2
  Interventions: Drug: Tremelimumab; Drug: Durvalumab; Radiation: Radiation

INTERVENTIONS:
Drug: Tremelimumab — Tremelimumab target the cancerous proteins and stop the cancer cells from suppressing the immune system
Drug: Durvalumab — Durvalumab target the cancerous proteins and stop the cancer cells from suppressing the immune system
  Other Names: Imfinzi
Radiation: Radiation — Radiation therapy is used to shrink cancer cells.

SUMMARY:
This research study is studying a combination of drugs as a possible treatment for Hepatocellular Carcinoma or Biliary Tract Cancer.

The interventions involved in this study are:

* Durvalumab
* Tremelimumab
* Radiation Therapy

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of investigational drugs to learn whether the drugs work in treating a specific disease. "Investigational" means that the drugs are being studied.

The FDA (the U.S. Food and Drug Administration) has not approved durvalumab for this specific disease but it has been approved for other uses.

The FDA has not approved tremelimumab as a treatment for any disease.

Both durvalumab and tremelimumab are antibodies (proteins that work with the immune system) that target proteins produced by the cancer cells. These cancerous proteins suppress the immune system which allows the cancer cells to grow. The study drugs may target these cancerous proteins and stop the cancer cells from suppressing the immune system.

The investigators hope that the combination of these study drugs with radiation therapy will help stop the cancer cells from growing and spreading.

ELIGIBILITY:
**After activation of a protocol amendment on July 14, 2022, only participants with biliary tract cancer will be permitted to enroll.**

Inclusion Criteria:

* Histologically or cytologically confirmed hepatocellular carcinoma or biliary tract cancer
* Locally advanced/unresectable or metastatic disease
* Age ≥ 18 years at time of study entry
* ECOG Performance Status ≤ 1
* One previously unirradiated lesion amenable to 8 Gy x 3 radiotherapy based on dosimetric organ tolerance AND another unirradiated measurable lesion (per irRECIST) outside of the radiation field
* Immunotherapy-naïve
* Progressed on, be intolerant of, or refused sorafenib [for HCC], second line treatment and beyond for cholangiocarcinoma or gemcitabine-based chemotherapy for biliary tract cancer
* The benefits of sorafenib have been discussed with the patient and the patient has refused treatment with sorafenib.
* Viral status (Hepatitis B and C) must be known. All HBV-positive patients must be on antiviral medication for viral suppression.

  * Patients with concomitant HBV infection must have a confirmed diagnosis of HBV characterized by the presence of hepatitis B core antibodies, and be sufficiently suppressed with active antiviral treatment (per local institutional practice) prior to enrollment to ensure adequate viral suppression (HBV deoxyribonucleic acid [DNA] <2000 IU/mL).
  * Patients with concomitant HCV infection must have confirmed diagnosis of HCV characterized by the presence of detectable HCV ribonucleic acid (RNA or anti-HCV antibody upon enrollment.
* Body weight ≥ 30 kg
* Child-Pugh Score of A. A score of B7 is allowed without severe ascites or without hepatic encephalopathy.
* Adequate organ and marrow function, defined as:

  * Hemoglobin ≥ 9 g/dL
  * ANC ≥ 1.5 x 10^9/L
  * Platelet count ≥75×109/L
  * Serum bilirubin ≤2.0× the upper limit of normal (ULN).
  * ALT and AST ≤ 3 x institutional ULN
  * Albumin > 2.8 g/dL
  * INR < 2.0
  * Calculated creatinine clearance > 40 mL/min as determined by Cockcroft-Gault (using actual body weight)
* Males:

  --Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)
* Females:

  --Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
* Ability to understand and the willingness to sign a written informed consent document
* Female subjects must be either of non-reproductive potential (i.e., post-menopausal by history: ≥ 50 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
* Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations with follow up

Exclusion Criteria:

* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
* Prior irradiation to the planned radiation target lesion
* Prior immunotherapy including but not limited to anti-CTLA4, including tremelimumab anti-PD-1, and anti-PD-L1, including durvalumab
* Concurrent enrollment in another study unless it is an observational (e.g. non-interventional) study
* Received live attenuated vaccines within 30 days of first dose
* Mean QT interval corrected for heart rate (QTc) ≥ 470 ms using Fredericia's Correction
* History of primary immunodeficiency
* History of solid organ transplantation
* Active or prior documented autoimmune disease within the past 2 years (NOTE: The following are exceptions to this criterion: Participants with vitiligo or alopecia; Participants with hypothyroidism (e.g. following Hashimoto syndrome) who are stable on hormone replacement; Participants with celiac disease controlled by diet alone: Participants with Grave's disease, or any chronic skin condition not requiring systemic treatment. Participants without active disease in the last 5 years may be included but only after consultation with the study physician.)
* Active or prior documented inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis)
* Prior other malignancy within 2 years (except for in situ disease, which is permissible)
* History of hypersensitivity to durvalumab, tremelimumab or any excipient
* History of (non-infectious) pneumonitis that required steroids; or evidence of interstitial lung disease or active, non-infectious pneumonitis
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses, or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Current or prior use of immunosuppressive medication within 28 days before the first dose of treatment on this protocol, with the exceptions of

  * Intranasal and inhaled corticosteroids
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent
  * Premedication for hypersensitivity reactions (e.g. to CT contrast for scans)
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Subjects with uncontrolled seizures
* Female subjects who are pregnant or breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period.
* Any unresolved toxicity NCI CTCAE Grade ≥ 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
* Patients with Grade ≥ 2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.

  --Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
* Brain metastases or spinal cord compression. Patients with suspected brain metastases at screening should have an MRI (preferred) or CT each preferably with IV contrast of the brain prior to study entry or brain metastases or spinal cord compression unless the patient is stable (asymptomatic; no evidence of new or emerging brain metastases; and stable and off steroids and anti-convulsants for at least 14-28 days prior to start of study treatment). Following radiotherapy and/or surgery of the brain metastases patients must wait 4 weeks following the intervention to confirm stability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-05-14 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Best Overall Response rate | Start of cycle 3, start of cycle 5, and then the start of every subsequent cycle for the remainder of treatment. One cycle is 4 weeks. (approximately 3 years)
  The number of participants that achieve either a complete response or partial response. Response rate (ORR) is assessed using irRECIST (Immune-related Response Evaluation Criteria In Solid Tumors). Response is evaluated with the use of computed tomography (CT) and magnetic resonance imaging (MRI) scans. Participants are evaluated for response for the duration of treatment.Treatment continues until disease progression, treatment is considered a safety risk, physicians decision, withdrawal from the study, or until the participant is lost to follow up. The best overall response recorded for each participant is reported.
  * Complete Response: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm (the sum may not be "0" if there are target nodes)
  * Partial Response: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters

SECONDARY OUTCOMES:
Number of Participants With Treatment Related Adverse Events | From the start of treatment until 30 days after the last dose of study drug is received (approximately 5 years)
  The number of participants that experience treatment related adverse events as assessed using Common Terminology Criteria for Adverse Events (CTCAE 4). Participants are evaluated for adverse events for the duration of treatment.Treatment continues until disease progression, treatment is considered a safety risk, physicians decision, withdrawal from the study, or until the participant is lost to follow up.
Overall Survival | From the start of treatment until the time of death or loss to follow-up (approximately 7 years)
  The median overall duration of survival as measured from the start of treatment until the time of death due to any cause or until the participant is lost to follow-up.
Disease Control Rate | Screening, start of cycle 3, start of cycle 5, and then the start of every subsequent 4-week cycle for the remainder of treatment (approximately 3 years)
  The number of participants that achieve a complete response (CR), partial response (PR), or stable disease (SD) as their best overall response as evaluated using irRECIST (Immune-related Response Evaluation Criteria In Solid Tumors). Participants are evaluated for response for the duration of treatment. Treatment continues until disease progression, treatment is considered a safety risk, physicians decision, withdrawal from the study, or until the participant is lost to follow up.
  * CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm (the sum may not be "0" if there are target nodes)
  * PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters
  * SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum of diameters while on study
Progression Free Survival | From the start of treatment until the time of death or loss to follow-up, whichever occurs first (approximately 7 years)
  The median amount of time from the start of treatment until the the first documentation of radiographic disease progression (per irRECIST) or death due to any cause, whichever occurs first. Participants who are alive with no documented disease progression by the data cutoff date for progression free survival analysis will be censored at the date of their last evaluable disease assessment.
  • Prior Progressive Disease: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: The appearance of one or more new lesions may be considered progression.)
Duration of Response | From first documentation of response to treatment until the time of disease progression (approximately 2 years)
  The median duration of time from first documentation of objective response to the first documented disease progression (per irRECIST). For participants who are alive and no documented progressive disease at the time of data cutoff for analysis, duration of response will be censored at the last evaluable disease assessment date.
Time to Disease Progression | From the start of treatment until the time of disease progression (approximately 7 years)
  The median duration of time from the start of treatment to the first documentation of radiographic disease progression (perirRECIST). Participants with no documented progressive disease by the data cutoff date for time to progression analysis will be censored at the date of their last evaluable disease assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore S. Hong, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No